CLINICAL TRIAL: NCT07309406
Title: Evaluating the Effects of a Nurse-Led Multicomponent Environmental Intervention on Stress Perception and Sleep Quality in ICU Patients: A Quasi-Experimental Study
Brief Title: Effect of a Nurse-Led Environmental Stressor Reduction Package on Perceived Stress and Sleep Quality in Intensive Care Unit Patients
Acronym: ICU-SLEEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, öznur balkan, Research Assistant, Fenerbahce University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FenerbahceU-ICUREST-2025
Record Dates: First submitted 2025-09-26; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sleep Disturbance
Keywords: Critical Care Nursing; Environmental Stressors; Intensive Care Unit; Sleep Quality; Quiet Night Protocol
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Masking Description: No parties are masked in this trial. The intervention (environmental stressor reduction package, including noise and light adjustment, eye mask use, and night-time care regulation) is directly observable by patients and healthcare providers. Therefore, participants, care providers, and outcome assessors are aware of group assignments. Data entry and statistical analyses will be performed independently to reduce potential bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quiet Night Protocol (Environmental Stressor Reduction Package) (Experimental): This arm will receive the Environmental Stressor Reduction Package, a multi-component nursing intervention designed to reduce environmental stressors in the ICU. The package includes:
  Noise control (≤45 dB, alarms adjusted, staff reminders)
  Circadian lighting adjustments (bedside lights off during sleep hours, local lighting for procedures, use of eye masks when appropriate)
  Thermal comfort monitoring (timpanically measured, blankets or controlled bedside warmers if needed)
  Restricted visitor traffic (no visitors after 22:00, quiet medical rounds at night)
  Adjustment of care activities (minimizing unnecessary night interventions, clustering nursing care before 22:00)
  Use of the "Quiet Night Checklist" by nurses at 22:00, 02:00, and 06:00 to standardize monitoring.
  Interventions: Behavioral: Environmental Stressor Reduction Package
- Standard ICU Care (No Intervention): This arm will receive routine ICU care without the structured Environmental Stressor Reduction Package. Standard care includes typical ICU monitoring, treatments, and nursing interventions according to hospital policies, without specific modifications for noise, light, thermal comfort, or visitor regulation beyond institutional standards.

INTERVENTIONS:
Behavioral: Environmental Stressor Reduction Package — A structured, nurse-led protocol implemented in the ICU to reduce environmental stressors that negatively affect patients' sleep quality. It combines noise reduction, circadian lighting adjustment, thermal comfort, visitor traffic regulation, and adjustment of care activities. Nurses use a standardized checklist ("Quiet Night Checklist") at three time points (22:00, 02:00, and 06:00) to ensure consistency and adherence.
  Arms: Quiet Night Protocol (Environmental Stressor Reduction Package)

SUMMARY:
This study aims to evaluate the effectiveness of a nurse-led "Environmental Stressor Reduction Package" on critically ill patients' perception of environmental stress and their sleep quality in the intensive care unit (ICU).

The package includes multi-component interventions such as reducing noise levels, adjusting lighting according to circadian rhythm, maintaining thermal comfort, limiting visitor traffic at night, and organizing nursing care to minimize sleep disruption. A structured "Quiet Night Checklist" will be used to monitor the implementation of these interventions during night shifts.

The study will be conducted in the 10-bed anesthesia and reanimation intensive care unit of Ümraniye Training and Research Hospital, İstanbul. Eligible adult patients who are awake, not under sedation, and able to communicate will be recruited. Participants in the intervention group will receive the Environmental Stressor Reduction Package for at least two and up to five consecutive nights, while the control group will continue to receive standard ICU care.

Outcomes will be measured using two validated tools:

The Intensive Care Unit Environmental Stressor Scale (ICUESS) to assess perceived environmental stress.

The Richards-Campbell Sleep Questionnaire (RCSQ) to evaluate self-reported sleep quality.

The findings of this study are expected to contribute to evidence-based nursing interventions in the ICU setting, by improving patients' sleep quality and reducing stressors associated with the intensive care environment.

DETAILED DESCRIPTION:
This semi-experimental study is designed to investigate the effect of a nurse-led "Environmental Stressor Reduction Package" on patients' perception of environmental stress and their sleep quality in the intensive care unit (ICU).

The intervention package includes five core components:

Noise control: Environmental sound levels will be maintained at ≤45 dB during night hours using a portable sound level meter (Benetech GM1351). Non-critical alarms will be silenced or reduced by 50%, and staff will be reminded to minimize unnecessary conversations at the bedside.

Lighting adjustment: Circadian rhythm-oriented lighting will be supported by turning off unnecessary bedside lights during sleep periods, using curtains to block external light, and providing patients with eye masks when needed.

Thermal comfort: As central air conditioning cannot be individually adjusted, tympanic temperature will be monitored and blankets or portable warmers will be used to ensure comfort.

Visitor regulation: No visitors will be allowed after 22:00, and physicians' or staff communications will be conducted as quietly as possible during patients' rest periods.

Nursing care organization: Routine nursing interventions such as hygiene care or repositioning will be scheduled before 22:00 whenever feasible, to minimize sleep interruption between 22:00 and 06:00.

The structured "Quiet Night Checklist" developed by the research team will be used to monitor the fidelity of the intervention. The checklist will be completed at 22:00, 02:00, and 06:00, covering all intervention domains. Each item is scored on a 3-point Likert scale (1 = not implemented, 2 = partially implemented, 3 = fully implemented).

Data collection will be carried out over a minimum of two and up to five consecutive nights of ICU stay, depending on patients' clinical course. The intervention group will receive the package, while the control group will continue to receive standard ICU care.

The primary outcome will be the change in patients' perceived environmental stress, measured by the Intensive Care Unit Environmental Stressor Scale (ICUESS), a validated 42-item instrument. The secondary outcome will be self-reported sleep quality, measured by the Richards-Campbell Sleep Questionnaire (RCSQ), a validated 5-item visual analogue scale. Both instruments have validated Turkish versions (Toptas et al., 2018; Demir et al., 2021).

It is anticipated that the intervention will reduce patients' stress perception and improve sleep quality compared to standard care. The findings will contribute to evidence-based nursing practices in ICU environments, highlighting the role of structured, nurse-led environmental modifications in improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older

Patients admitted to the intensive care unit (ICU)

Awake and able to communicate (not under sedation or mechanical ventilation)

Expected to remain in the ICU for at least 2 consecutive nights

Voluntary participation with written informed consent

Exclusion Criteria:

* Patients under 18 years old

Patients diagnosed with delirium or severe cognitive impairment

Patients with a history of psychiatric illness affecting sleep or stress perception

Patients under continuous sedative or opioid infusion

Patients discharged from the ICU or deceased before completing the intervention period (2-5 nights)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in environmental stress perception | Baseline and Day 5
  Environmental stress perception will be assessed using the Intensive Care Unit Environmental Stressor Scale (ICUESS), Turkish validated version (Toptaş, Yıldız, & Khorshid, 2018). The ICUESS consists of 42 items rated on a 4-point Likert scale ranging from 0 (not stressful) to 3 (very stressful), yielding a total score range of 0 to 126. Higher total scores indicate greater perceived environmental stress.

SECONDARY OUTCOMES:
Change in sleep quality | Baseline and Day 5
  Sleep quality will be assessed using the Richards-Campbell Sleep Questionnaire (RCSQ), Turkish validated version (Demir, Zaybak, & Erdoğan, 2021). The RCSQ consists of 5 items rated on a visual analog scale ranging from 0 to 100 mm. The total score is calculated as the mean of the five items, yielding a score range of 0 to 100. Higher scores indicate better subjective sleep quality.
Correlation between environmental stress perception and sleep quality | Day 5 (end of intervention)
  The association between ICUESS total scores and RCSQ mean scores will be analyzed to determine the relationship between perceived environmental stressors and subjective sleep quality.

OTHER OUTCOMES:
Intervention adherence (implementation fidelity) | Nightly, at 22:00, 02:00, and 06:00 during intervention nights (2-5 nights).
  Adherence to the Quiet Night Protocol will be evaluated using the Sessiz Gece Kontrol Listesi (Quiet Night Control Checklist), developed by the research team. Items are scored with a 3-point Likert scale (1 = not applied, 2 = partially applied, 3 = fully applied). Higher total scores indicate higher fidelity of protocol implementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
What data will be shared? Anonymized individual participant data (IPD) including demographic information (age, sex, diagnosis, length of ICU stay) and primary outcome measures (ICUESS scores and RCSQ scores). No identifying information (e.g., names, contact details, medical record numbers) will be shared.
  When will data be available? De-identified data will be available beginning 6 months after publication of the main study results and will remain accessible for 2 years.
  With whom and under what conditions? Data will be shared with academic researchers upon submission of a methodologically sound proposal and approval from an institutional review board (IRB) or ethics committee. Interested researchers must sign a data-sharing agreement to ensure confidentiality and appropriate use of data.
  How will data be shared? Data will be provided through secure, password-protected institutional servers. Requests can be directed to the principal investigator via email.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Individual participant data (IPD) and supporting documents will be available beginning 6 months after publication of the primary results and will remain accessible for a period of 2 years.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan, informed consent form, and analytic code) will be made available to qualified researchers. Access will be granted only to investigators affiliated with academic or health research institutions who provide a methodologically sound research proposal and obtain local ethics approval. Researchers must sign a data use agreement to ensure data security and confidentiality. Access will be provided through secure, password-protected electronic transfer upon request to the study sponsor.